CLINICAL TRIAL: NCT04012645
Title: A Study Assessing Perfusion Outcomes With Near Infrared-Indocyanine Green Imaging System in Laparoscopic Total Mesorectal Excision for Mid- or Low-rectal CanceR
Brief Title: Perfusion Outcomes With Near Infrared-Indocyanine Green Imaging System in Laparoscopic Total Mesorectal Excision for Mid- or Low-rectal CanceR
Acronym: POSTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongtao Zhang (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Chao Yang Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Chinese PLA General Hospital (Other); Peking University People's Hospital (Other); Peking University Cancer Hospital & Institute (Other); Beijing Hospital (Other Government); Changhai Hospital (Other); Ruijin Hospital (Other); RenJi Hospital (Other); Fudan University (Other); Guangdong Provincial People's Hospital (Other); Southern Medical University, China (Other); First Hospital of China Medical University (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Zhongtao Zhang, Director of General Surgery of Beijing Friendship Hospital, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Poster
Record Dates: First submitted 2019-07-06; First posted 2019-07-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms
Keywords: Rectal Neoplasms; Indocyanine Green; Anastomotic Leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Underwent laparoscopic TME and colon-rectum or colon-anal anastomosis. near infrared-indocyanine green imaging system was used during the surgeries.
  Interventions: Procedure: application of near infrared-indocyanine green imaging system
- control group (Active Comparator): Underwent laparoscopic TME operation, and the operator judged anastomotic blood supply with naked eyes and performed the surgical intervention based on the experience
  Interventions: Procedure: Non-application of near infrared-indocyanine green imaging system

INTERVENTIONS:
Procedure: application of near infrared-indocyanine green imaging system — Underwent laparoscopic TME and colon-rectum or colon-anal anastomosis. near infrared-indocyanine green imaging system was used to evaluate the anastomotic flood perfusion during the operation; The operator may decide whether to change the surgical programme based on the outcome of the evaluation.
  Arms: experimental group
Procedure: Non-application of near infrared-indocyanine green imaging system — Underwent laparoscopic TME operation, and the operator judged anastomotic blood supply with naked eyes and performed the surgical intervention based on the experience
  Arms: control group

SUMMARY:
It is a multicenter, prospective, and randomized controlled clinical study of patients with mid- or low- rectal cancer who received laparoscopic TME surgery aims to explore whether the application of near infrared-indocyanine green imaging system can evaluate the anastomotic blood perfusion accurately, and optimize the surgical procedures, or even reduce the incidence rates of postoperative anastomotic leakage in mid- or low- rectal cancer patients.

DETAILED DESCRIPTION:
In total mesorectal excision of rectal cancer, accurate assessment of rectal anastomotic blood supply is crucial: for insufficient anastomotic blood supply is an important cause of postoperative anastomotic leakage, and once anastomotic leakage occurs, the perioperative mortality rate of patients is reportedly 16%. In the past, the assessment of anastomotic blood supply mainly depended on the experience of the surgeon and lacked objective and accurate assessment methods. In recent years, the application of near-infrared fluorescence laparoscopic imaging technology has provided a new way to accurately evaluate anastomotic perfusion. At present, the technology has been applied to evaluate anastomotic blood supply in colorectal cancer surgery worldwide, and its safety and reliability have been confirmed. However, whether the application of this technology can reduce the incidence of anastomotic leakage after total mesorectal excision for rectal cancer and thus benefit patients still needs high-level evidence-based medical evidence support with multi-centers and large samples.Thus, a multicenter, prospective, and randomized controlled clinical study of patients with mid- or low- rectal cancer who received laparoscopic TME surgery was intend to conduct to explore whether the application of near infrared-indocyanine green imaging system can evaluate the anastomotic blood perfusion accurately, and optimize the surgical procedures, or even reduce the incidence rates of postoperative anastomotic leakage in mid- or low- rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* The age was over 18 years at the time of diagnosis;
* Diagnosis of rectal carcinoma and was confirmed by preoperative pathology;
* MRI was performed before operation, and the distance between the lower margin of tumor and the anal margin was no more than 10cm;
* The colon-rectum or colon-anus anastomosis was performed by laparoscopic TME operation
* The "spleen area" was not free during the operation
* Baseline clinical tumor stage TNM Ⅰ-Ⅲ phase: cT1-4N0-2M0 （AJCC-8 version）;

Exclusion Criteria:

* Allergic to ICG or iodine;
* Patients with intestinal obstruction, intestinal perforation, intestinal bleeding who need emergency operation;
* Patients requiring combined organ resection that the tumor involves adjacent organs;
* Patients with recurrence of tumor or distant metastasis;
* Patients with multiple colorectal cancer;
* Patients with history of inflammatory bowel disease or familial adenomatous polyposis;
* Patients who have participated in or are participating in other clinical trials in the past four weeks;
* Patients that ASA level is larger than III;
* Physical condition: Patients with KPS less than or equal to 60 points or ECOG larger than or equal to 2 points;
* Patients with hepatic dysfunction and MELD larger than 12 points;
* Patients with a history of serious mental illness;
* Pregnant or lactating women;
* Patients who are improper to participate in the study in the opinion of the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage | within 30 days after operation
  Anastomotic leakage occured within 30 days after operation. The diagnostic criteria for AL include: Flow of gas, abscess, or excrement from pelvic drainage tube, surgical incision or vagina; Accompanied by fever, peritonitis and other systemic symptoms; And AL confirmed by digestive tract radiography, CT scan or enteroscopy.

SECONDARY OUTCOMES:
the change of surgical precedure | within the operation time
  the change of intraoperative decision, including: (1) The change of the position of intestinal dissection; (2) Anastomotic stoma was removed and rebuilt or re-performed hartmann operation; (3) The performance of unplanned, preventive orifice, etc. due to ICG test results.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Professor, Principal Investigator — Beijing Friendship Hospital
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital medical University, Beijing, Xicheng Dis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun L, Gao J, Wu G, Meng C, Yang Z, Wei P, Yao H, Zhang Z. Perfusion outcomes with near-infrared indocyanine green imaging system in laparoscopic total mesorectal excision for mid-rectal or low-rectal cancer (POSTER): a study protocol. BMJ Open. 2024 May 9;14(5):e079858. doi: 10.1136/bmjopen-2023-079858. PMID 38724058